CLINICAL TRIAL: NCT03729453
Title: Intra-operative Pancreatoscopy in Patients With Intraductal Papillary Mucinous Neoplasm (IPMN)
Brief Title: Intra-operative Pancreatoscopy in Patients With IPMN
Status: Active, not recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: E7107
Record Dates: First submitted 2018-11-01; First posted 2018-11-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Intraductal Papillary Mucinous Neoplasm
Keywords: IPMN; SpyGlass; Pancreatoscopy; Intraductal Papillary Mucinous Neoplasm; Intraoperative; Surgical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Intraoperative Pancreatoscopy: All subjects will undergo the intraoperative pancreatoscopy with SpyGlass procedure.
  Interventions: Device: SpyGlass

INTERVENTIONS:
Device: SpyGlass — Visualization of main pancreatic duct with SpyGlass catheter.

SUMMARY:
To demonstrate the added value of intraoperative pancreatoscopy in patients undergoing partial pancreatic resection for the treatment of Intraductal Papillary Mucinous Neoplasm (IPMN) as it pertains to detection of discontinuous (skip) lesions in the remnant pancreas; to generate a hypothesis for a subsequent randomized control trial.

DETAILED DESCRIPTION:
The primary objective of this study is to demonstrate the added value of intraoperative pancreatoscopy in patients undergoing partial pancreatic resection for the treatment of Intraductal Papillary Mucinous Neoplasm (IPMN) as it pertains to detection of discontinuous (skip) lesions in the remnant pancreas. A secondary study objective is to generate a hypothesis for a subsequent randomized controlled trial comparing diagnostic accuracy of intra-operative pancreatoscopy and SpyBite™ with the diagnostic accuracy of intra-operative frozen section in patients undergoing resection

ELIGIBILITY:
Inclusion Criteria:

1. Patient scheduled for surgery for suspected MD-IPMN or Mixed IPMN within 4-6 weeks of enrollment
2. Diameter of pancreatic main duct >5mm on pre-operative MRI or CT
3. Written informed consent from patient to participate in the study, including compliance with study procedures

Exclusion Criteria:

1. Contraindication for pancreatoscopy
2. Age: less than 18 years
3. Pregnant women, evaluated per local clinical standard

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for surgery for suspected MD-IPMN or Mixed IPMN resection.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Rate of detection of discontinuous (skip) lesions along the main pancreatic duct | During index procedure
  Rate of detection of discontinuous (skip) lesions along the main pancreatic duct of patients with IPMN using intraoperative pancreatoscopy based on visual impression of IPMN and/or pancreatoscopy guided biopsies

SECONDARY OUTCOMES:
Technical success | During index procedure
  Ability to advance the pancreatoscope along the entire main pancreatic duct length or until clinically needed; to visualize the potential lesion(s); or to obtain a tissue sample with SpyBite where applicable
Adverse Event Evaluation | Five years
  Evaluate all serious adverse events related to the intraoperative pancreatoscopy procedure and/or device
Recurrence | Five years
  Recurrence of IPMN within 5 years post-surgery evaluated with regular MRI or alternative radiological method
Comparison of visual and biopsy diagnosis | During index procedure
  Comparison based on exploration with Spy Glass of the resected specimen
Inter-observer correspondence of visual impression of IPMN | During index procedure
  Based on intra-operative impression and on review of recorded pancreatoscopy images/videos

CONTACTS AND LOCATIONS:
Overall Officials: Marco Del Chiaro, MD, Principal Investigator — University of Colorado, Denver; G.V. Rao, MD, Principal Investigator — Asian Institute of Gastroenterology; Richard Burkhart, MD, Principal Investigator — Johns Hopkins University; Marc Besselink, MD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Yi Miao, MD, Principal Investigator — Nanjing Medical University; Sohei Satoi, MD, Principal Investigator — Kansai Medical University; Urban Arnelo, MD, Principal Investigator — University Hospital, Umeå; Christian Schmidt, MD, Principal Investigator — Indiana University Health
Locations (8):
- United States (3):
  - University of Colorado Hospital, Denver, Colorado
  - Indiana University Health, Indianapolis, Indiana
  - Johns Hopkins Hospital University, Baltimore, Maryland
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, China
- Asian Institute of Gastroenterology, Hyderabad, India
- Kansai Medical University, Hirakata, Osaka, Japan
- Academic Medical Center, Amsterdam, Netherlands
- University Hospital of UMEA, Umeå, Sweden

REFERENCES:
- [Derived] Grewal M, Habib JR, Paluszek O, Cohen SM, Wolfgang CL, Javed AA. The Role of Intraoperative Pancreatoscopy in the Surgical Management of Intraductal Papillary Mucinous Neoplasms: A Scoping Review. Pancreas. 2024 Mar 1;53(3):e280-e287. doi: 10.1097/MPA.0000000000002294. Epub 2024 Jan 26. PMID 38277399